CLINICAL TRIAL: NCT02139163
Title: Epidemiological Study on Community Acquired Pneumonia
Acronym: CAPNETZ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: U1111-1147-8393
Record Dates: First submitted 2014-01-24; First posted 2014-05-15 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Community Acquired Pneumonia
Keywords: Community acquired pneumonia; CAP; CAPNETZ; age ≥18; infiltrate on chest X-ray; cough or production of purulent sputum; pathologic lung auscultation; fever
MeSH Terms: conditions — Community-Acquired Pneumonia; Cough; Fever | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with pneumonia
  Interventions: Other: Cohort Study

INTERVENTIONS:
Other: Cohort Study

SUMMARY:
Long-term objectives of the basic research part are improvement of CAP-management with respect to therapy, diagnosis and prevention to contribute to a better care of patients with pneumonia.

DETAILED DESCRIPTION:
Long-term objectives of the basic research part are improvement of CAP-management with respect to therapy, diagnosis and prevention to contribute to a better care of patients with pneumonia. The aim of the study CAPNETZ is to improve diagnosis, treatment and patient care.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* infiltrate on chest X-ray
* further Inclusion criteria: cough or production of purulent sputum or pathologic lung auscultation (crackles) or fever

Exclusion Criteria:

* hospital inpatient treatment within the last 28 days
* Immune suppressed patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 10150 (Estimated)
Dates: Start 2002-10; Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
diagnosis | 2 weeks
  Assessment of diagnosis:
  Patients will be asked for example, about their diagnosis, comorbidities, specific risk factors and pneumonia symptoms.
therapy | 2 weeks
  Assessment of therapy:
  Patients will be asked about their therapy due to pneumonia symptoms, previous therapy, medication History etc.
hospitalization | 2 weeks
  Assessment of hospitalization:
  Patients will be asked about hospitalization, date, time and duration of hospitalization due to pneumonia symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Welte, Prof. Dr., Study Chair — Hannover Medical School
Locations (2):
- Germany (2):
  - CAPNETZ FOUNDATION Hannover Medical School (MHH), Hanover, Lower Saxony
  - Hannover Medical School, Hanover, Lower Saxony

REFERENCES:
- [Result] Zobel K, Martus P, Pletz MW, Ewig S, Prediger M, Welte T, Buhling F; CAPNETZ study group. Interleukin 6, lipopolysaccharide-binding protein and interleukin 10 in the prediction of risk and etiologic patterns in patients with community-acquired pneumonia: results from the German competence network CAPNETZ. BMC Pulm Med. 2012 Feb 20;12:6. doi: 10.1186/1471-2466-12-6. PMID 22348735
- [Result] Klapdor B, Ewig S, Schaberg T, Rohde G, Pletz MW, Schutte H, Welte T; CAPNETZ study group. Presentation, etiology and outcome of pneumonia in younger nursing home residents. J Infect. 2012 Jul;65(1):32-8. doi: 10.1016/j.jinf.2012.02.003. Epub 2012 Feb 10. PMID 22330772
- [Result] Lepper PM, Ott S, Nuesch E, von Eynatten M, Schumann C, Pletz MW, Mealing NM, Welte T, Bauer TT, Suttorp N, Juni P, Bals R, Rohde G; German Community Acquired Pneumonia Competence Network. Serum glucose levels for predicting death in patients admitted to hospital for community acquired pneumonia: prospective cohort study. BMJ. 2012 May 28;344:e3397. doi: 10.1136/bmj.e3397. PMID 22645184
- [Result] Kolditz M, Hoffken G, Martus P, Rohde G, Schutte H, Bals R, Suttorp N, Pletz MW; CAPNETZ study group. Serum cortisol predicts death and critical disease independently of CRB-65 score in community-acquired pneumonia: a prospective observational cohort study. BMC Infect Dis. 2012 Apr 13;12:90. doi: 10.1186/1471-2334-12-90. PMID 22501026
- [Result] Klapdor B, Ewig S, Pletz MW, Rohde G, Schutte H, Schaberg T, Welte T; CAPNETZ Study Group. Community-acquired pneumonia in younger patients is an entity on its own. Eur Respir J. 2012 May;39(5):1156-61. doi: 10.1183/09031936.00110911. Epub 2011 Nov 16. PMID 22088967
- [Result] Ewig S, Klapdor B, Pletz MW, Rohde G, Schutte H, Schaberg T, Bauer TT, Welte T; CAPNETZ study group. Nursing-home-acquired pneumonia in Germany: an 8-year prospective multicentre study. Thorax. 2012 Feb;67(2):132-8. doi: 10.1136/thoraxjnl-2011-200630. Epub 2011 Nov 5. PMID 22058186
- [Derived] Glockner V, Pletz MW, Rohde G, Rupp J, Witzenrath M, Barten-Neiner G, Kolditz M; CAPNETZ Study Group. Early post-discharge mortality in CAP: frequency, risk factors and a prediction tool. Eur J Clin Microbiol Infect Dis. 2022 Apr;41(4):621-630. doi: 10.1007/s10096-022-04416-5. Epub 2022 Feb 8. PMID 35137301